CLINICAL TRIAL: NCT00729092
Title: Additional (Positron Emission Tomography)PET Scan of Brain in Patients Undergoing PET Scan for Diseases Unrelated to Brain
Brief Title: Additional Positron Emission Tomography (PET) Scan of Brain in Patients Undergoing PET Scan for Diseases Unrelated to Brain
Status: Completed | Type: Observational
Sponsor: Asokumar Buvanendran (Other)
Responsible Party: Sponsor-Investigator, Asokumar Buvanendran, Attending Physician, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Other Study IDs: 08042105
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Pain
Keywords: PET SCAN; PAIN LEVELS
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific Aims:

• The primary objective is to delineate the brain structures that are involved in pain using Positron Emission Tomography (PET) imaging.

Hypothesis:

Pain will result in increases in metabolism and neuronal activity in specific delineated areas of the brain.

DETAILED DESCRIPTION:
Background and Significance:

Despite advancement in pain management, pain relief and patient satisfaction are still inadequate in many patients. Functional imaging techniques have recently made it possible to identify the main cerebral components of the human nociceptive system. These comprise at least two main human nociceptive components working in parallel called the medial and lateral pain systems. This has provided a physical construct for the concept of the human pain matrix. Careful study of these areas of the human brain has the potential to drive development of new classes of analgesic compounds. PET is an imaging technique that can quantify increases in nerve cell activity in selective regions of the brain (1-5). PET provides the means to measure tissue concentrations of labeled drugs in brain and other tissues and also to measure changes in receptor occupancy.

Earlier studies have examined the pattern of increased brain activity that follows experimentally-induced acute pain (2) and chronic pain syndromes (1,3,5). Distal pain pathways (e.g. spinothalamic tract) project to the thalamus and then discrete regions of the cortex via thalamocortical projections. Among cortical areas involved in sensation, perception, and attention in both humans and monkeys are anterior cingulate gyrus, insular cortex, primary somatosensory cortex, and secondary somatosensory cortex. PET studies with experimental human pain also demonstrate activation in brain areas related to sensory-motor integration. However, depending on the type of noxious stimulation, different areas of brain are activated (2). Components of the lateral system such as the primary somatosensory (SI) cortex do appear to be frequently activated with tonic (non-phasic experimental pain) and phasic pain (67% and 69% of studies show activations, respectively). But only 23% of studies of chronic clinical pain studies demonstrate activation of SI.

We have performed the first clinical study (IRB study #05121504) to investigate the change in brain activity associated with significant postoperative pain (6). This was an IRB-approved study with just one patient to establish that the methods we have developed will be sensitive enough for a more complete randomized clinical trial. We determined that postsurgical pain is associated with increased activity in the contralateral primary somatosensory cortex. Other brain regions showing increased postsurgical activity were the contralateral parietal cortex, bilateral pulvinar and ipsilateral medial dorsal nucleus of the thalamus, contralateral putamen, contralateral superior temporal gyrus, ipsilateral fusiform gyrus, ipsilateral posterior lobe and contralateral anterior cerebellar lobe. We have received permission from the IRB to perform a larger study with 21 patients (IRB study #07050273).

Although fMRI has also been used for functional brain imaging, the advantages of PET over fMRI are (7):

PET is detected in neural tissue, while fMRI is detected in the venous compartment

1. PET with 18F-fluoro-2-deoxyglucose (FDG) gives a direct measure of glucose metabolism, while fMRI measures blood flow by measuring changes in deoxyhemoglobin concentration
2. PET has a larger signal-to-noise ratio than fMRI
3. PET is less susceptible to movement artifacts than fMRI
4. With PET for brain only the head is in the scanner, less claustrophobic than fMRI
5. PET does not have the inhomogeneity artifacts of fMRI
6. PET has the capacity for future ligand-binding studies (e.g. opioid receptor)

Comparable brain imaging studies have not been performed in primates due to the difficulty of having an animal not move for the duration of the scan, without the use of anesthetics.

To better interpret our PET brain images in the above clinical trials, we need more baseline data on the variability in brain activation from person-to person, especially in people with no or minimal pain. Clinical oncology utilizes PET imaging for the diagnosis and monitoring of many types of cancer, e.g. Hodgkin's disease, non-Hodgkin's lymphoma, and lung cancer. The brain of these individuals can be considered within normal range and could be a control for our other studies involving postoperative pain and its alleviation. To obtain these 'control' brain scans, a patient being scanned for diseases outside the brain would not have to have an additional radionuclide injection. Instead, after the primary body scan is completed, the patient platform would be moved slightly so the head is now centered in the scanner, and the scanning process resumed, for approximately 20 minutes. Since the half-life of the FDG radionuclide is about 110 min, there will still be adequate signal available to be picked up by the detector during this secondary scan.

ELIGIBILITY:
Inclusion Criteria:1.

* Subject who can understand and communicate in English

Exclusion Criteria:

* Younger than 18 years or older than 80 years.
* Greater than 90 kg body weight.
* American Society of Anesthesiologists physical status IV.
* Patient who is currently enrolled in another investigational study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between 18-80 years of age
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain Assessment Pain scores using the verbal rating scale, with 0 corresponding to "no pain" and 10 to the "worst imaginable pain" will be assessed prior to the primary PET scan | 20 mins

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States